CLINICAL TRIAL: NCT02688114
Title: Healing of the Esophageal Mucosa After Radiofrequency Ablation of Barrett's Esophagus
Brief Title: Healing of the Esophageal Mucosa After RFA of Barrett's Esophagus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dallas VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Stuart Spechler, Chief, Division of Gastroenterology, Dallas VA Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15-076
Record Dates: First submitted 2016-02-11; First posted 2016-02-23 (Estimated); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Barrett Esophagus
MeSH Terms: conditions — Barrett Esophagus | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Barrett's Esophagus Treatment (Experimental): All participants are in the treatment arm. Patients with Barrett's esophagus will undergo baseline surveillance endoscopy, be treated with radiofrequency ablation, and undergo follow up endoscopy 1, follow up endoscopy 2, and follow up endoscopy 3.
  Interventions: Procedure: Baseline surveillance endoscopy; Procedure: Radiofrequency ablation; Procedure: Follow up endoscopy 1; Procedure: Follow up endoscopy 2; Procedure: Follow up endoscopy 3

INTERVENTIONS:
Procedure: Baseline surveillance endoscopy — All study participants will undergo endoscopy with NinePoint NvisionVLE volumetric laser endomicroscopy and biopsy of the esophageal mucosa and gastric cardia.
Procedure: Radiofrequency ablation — All study participants will undergo radiofrequency ablation of Barrett's esophagus
Procedure: Follow up endoscopy 1 — All study participants will undergo follow up endoscopy 1 week after RFA, which includes endoscopy, NinePoint NvisionVLE volumetric laser endomicroscopy, and biopsies.
Procedure: Follow up endoscopy 2 — All study participants will undergo follow up endoscopy 2 weeks after RFA, which includes endoscopy, NinePoint NvisionVLE volumetric laser endomicroscopy, and biopsies.
Procedure: Follow up endoscopy 3 — All study participants will undergo follow up endoscopy 4 weeks after RFA, which includes endoscopy, NinePoint NvisionVLE volumetric laser endomicroscopy, and biopsies.

SUMMARY:
Radiofrequency ablation (RFA) is a mainstay of treatment for patients who have Barrett's esophagus (BE) with dysplasia. For unclear reasons, Barrett's esophagus recurs after successful RFA treatment in approximately 1/3 of patients. The aim of this study is to characterize the healing process of the esophageal mucosa, histologically and at the molecular level, after RFA for non-dysplastic and dysplastic Barrett's esophagus.

DETAILED DESCRIPTION:
Radiofrequency ablation (RFA) is a mainstay of treatment for patients who have Barrett's esophagus (BE) with dysplasia. For unclear reasons, Barrett's esophagus recurs after successful RFA treatment in approximately 1/3 of patients. Little is known of how the esophagus heals after RFA treatment, and a better understanding of this healing process might provide insights into how to prevent Barrett's metaplasia from recurring after successful ablation.

The aim of this study is to characterize the healing process of the esophageal mucosa, histologically and at the molecular level, after RFA for non-dysplastic and dysplastic Barrett's esophagus. Patients with Barrett's esophagus will undergo surveillance endoscopy with biopsy. This will be followed by RFA treatment of the BE and follow up endoscopy will be performed 1, 2, and 4 weeks after RFA. Healing at each time point will be assessed endoscopically, and molecular markers related to healing will be studied. Stem cell expression markers, immune cells and markers of epithelial-mesenchymal transition will be compared with baseline expression for each patient. Protocol has been modified to provide a collaborative effort between the Dallas VAMC and Baylor Scott & White Medical Center in Dallas, TX. Veteran participants electing to participate will receive initial screening and endoscopy at the Dallas VAMC and will continue with RFA and follow-up endoscopies at Baylor. An identical protocol has been approved at Baylor Scott & White Medical center. Patients who are screened and enrolled at Baylor will receive all treatments at that location.

ELIGIBILITY:
Inclusion Criteria:

- Barrett's esophagus

Exclusion Criteria:

* inability to provide informed consent
* esophageal varices
* treatment with warfarin
* coagulopathy that precludes safe biopsy of the esophagus (including platelet count <100,000/mm3, INR (international normalized ratio) >1.5)
* allergy to fluorescein sodium
* comorbidity that precludes safe participation in the study
* pregnancy or breastfeeding status

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2020-01-29 (Actual); Study Completion 2020-01-29 (Actual)

PRIMARY OUTCOMES:
Change in the Percent of Mucosa Healed by Neosquamous Epithelium | 1 week, 2 weeks, 4 weeks
  % of the esophageal mucosa healed by Neosquamous epithelium at 1 week, 2 weeks, and 4 weeks after RFA

SECONDARY OUTCOMES:
Change in expression of genes associated with epithelial-mesenchymal transition, stem cells, and submucosal glands | 1 week, 2 weeks, 4 weeks
  Measurement of gene expression in the esophageal mucosa 1 week, 2 weeks, 4 weeks after RFA. Genes related to the process of epithelial-mesenchymal transition, stem cells and submucosal glands will be studied.
Change in inflammatory cell infiltrate | 1 week, 2 weeks, 4 weeks
  Measurement of the changes in inflammatory cell infiltration (neutrophils, eosinophils, lymphocytes) of the esophageal mucosa 1 week, 2 weeks, and 4 weeks after RFA

CONTACTS AND LOCATIONS:
Overall Officials: Stuart J Spechler, MD, Principal Investigator — Baylor Scott and White Research Institute
Locations (2):
- United States (2):
  - Baylor Scott and White Research Institute, Dallas, Texas
  - Dallas VA Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No